CLINICAL TRIAL: NCT00691561
Title: Culturally-Tailored HIV Risk Reduction for African-American MSM (Project ABLE: African-Americans Building Life Empowerment
Brief Title: Culturally-Tailored HIV Risk Reduction for African-American MSM
Acronym: Project ABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Diverse and Resilient (Unknown); Charles D Productions (Unknown); Milwaukee LGBT Community Center (Other)
Responsible Party: David Seal, Principal Investigator, Medical College of Wisconsin- Center for AIDS Intervention Research
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-5394
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV Prevention; African American; Black; gay; Men who have sex men; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants receive HIV counseling and testing and 8 intervention sessions to assist them with reducing unsafe sexual behaviors.
  Interventions: Behavioral: Project ABLE
- 2 (No Intervention): Participants receive HIV counseling and testing only.

INTERVENTIONS:
Behavioral: Project ABLE — Participants will receive HIV counseling and testing. Those selected for the intervention arm will attend small groups consisting of 10 men who meet once a week for 8 consecutive weeks. The weekly two hour discussion sessions will address HIV risk behavior within a framework of contextual influences that may moderate men's risk reduction motivation and behavior. The factors include identity, stigma, connections to community, and situation factors.
  Arms: 1

SUMMARY:
The purpose of this study to conduct a small randomized control trial to compare the relative effectiveness of a single-session of HIV testing and counseling risk reduction intervention (HCT-only) to an enhanced intervention that includes the standard HCT intervention plus a theory-based and culturally-tailored group-level intervention designed to reduce or eliminate HIV and STI risk behaviors (HCT-plus) among African-American men who have sex with men (AA-MSM).

DETAILED DESCRIPTION:
The HCT-plus intervention will consist of the HCT-only intervention, as well as 8 small group intervention sessions focused on HIV risk reduction. Small groups will consist of 10 men who will meet once-a-week for 8 consecutive weeks. Each meeting will last approximately 2 hours. In each small group session, staff will work with men to reassess their HIV risk behavior, re-prioritize their goals as appropriate, and provide motivational support for their risk reduction accomplishments. Participants will be asked to discuss ways they have successfully avoided HIV risk behavior since the previous session, as well as to discuss situations in which they found it difficult to avoid risk. Staff will reinforce successful risk avoidance, and problem-solve with men to overcome barriers to risk reduction.

ELIGIBILITY:
Inclusion Criteria:

* reside in Milwaukee county;
* are at least 18 years of age;
* self-identify as male;
* self-identify as Black or African-American;
* can provide informed consent;
* report unprotected anal sex with a man in the past 3 months;
* report at least two sexual partners with whom they have had unprotected anal or vaginal sex in the past 3 months;
* are willing to be tested for HIV using rapid oral fluid procedures or willing to provide evidence of HIV seropositivity

Exclusion Criteria:

* Under 18 years of age,
* involvement in a HIV prevention study currently or in the past 6 months,
* Participation in the pilot phase

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The HCT-plus intervention will result in a greater proportion of men who abstain from anal and vaginal intercourse. | 3 months after completing intervention

SECONDARY OUTCOMES:
The HCT-plus intervention will result in a smaller proportion of men who had an act of anal or vaginal intercourse without the use of a condom. | 3 months after completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Seal, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Diverse and Resilient, Milwaukee, Wisconsin, United States